CLINICAL TRIAL: NCT04461015
Title: The Effect of the Interaction of Glucagon and Insulin on Endogenous Glucose Production in Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Vella (Other)
Responsible Party: Sponsor-Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-001570
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.4mU Insulin (Other): During the euglycemic clamp insulin will be infused at 0.4mU/Kg/Min
  Interventions: Drug: 0.4mU Insulin followed by withdrawal period followed by 0.8mU study; Drug: 0.8mU Insulin followed by withdrawal period followed by 0.4mU study
- 0.8mU Insulin (Other): During the euglycemic clamp insulin will be infused at 0.8mU/Kg/Min
  Interventions: Drug: 0.4mU Insulin followed by withdrawal period followed by 0.8mU study; Drug: 0.8mU Insulin followed by withdrawal period followed by 0.4mU study

INTERVENTIONS:
Drug: 0.4mU Insulin followed by withdrawal period followed by 0.8mU study — Clamp study with insulin infused at 0.4 mU/Kg/min, followed by a 2 week withdrawal period followed by a clamp study with insulin infused at 0.8 mU/Kg/min
  Other Names: 0.4 then 0.8
Drug: 0.8mU Insulin followed by withdrawal period followed by 0.4mU study — Clamp study with insulin infused at 0.8 mU/Kg/min, followed by a 2 week withdrawal period followed by a clamp study with insulin infused at 0.4 mU/Kg/min
  Other Names: 0.8 then 0.4

SUMMARY:
The purpose of this research is to help understand the relative importance of changes in insulin secretion (which lowers glucose) and changes in glucagon (which raises glucose) to regulate metabolism and the body's ability to make glucose.

DETAILED DESCRIPTION:
Study A (Insulin 0.4mU/Kg/min): Subjects will be admitted to the CRTU at approximately 1700 on the day prior to study. They will then consume a standard 10kcal/kg meal (55% carbohydrate, 30% fat, 15% protein, caffeine free) and fast overnight. Blood will then be sampled for baseline enrichment and 2H20 (1.67g/kg of body water) will be given in 3 divided doses at 2200, 2400 and 0200. The following morning (approximately 0530), a forearm vein will be cannulated to allow infusions to be performed. In addition, a cannula will be inserted retrogradely into a vein of the contra-lateral dorsum of the hand. This will be placed in a heated Plexiglas box maintained at around 120oF to allow sampling of arterialized venous blood. At approximately 0600 (-180 min), a primed, (10microCi prime, 0.1microCi/min continuous) infusion containing trace amounts of glucose labeled with [3-3H] glucose will be started and continued till 0900 (0 min).

At 0900 (0 min), the infusion will be varied so as to mimic the anticipated pattern of fall of EGP. In addition, glucose also labeled with [3-3H] glucose will be infused so as to maintain glucose concentrations at ~ 95mg/dL. Peripheral venous glucose concentrations will be measured every 10 minutes to allow the infusion rate of glucose to be adjusted as necessary.

Simultaneously, an infusion of somatostatin (60ng/kg/min) will be started at time 0 to inhibit endogenous islet secretion and therefore ensure identical portal insulin concentrations on the two study days. Insulin will be infused at a constant rate known to produce ~ 50% suppression of EGP (0.4mU/Kg/min).

From 0900 (0 min) to 1030 (90 min) no glucagon will be infused. Subsequently, a glucagon infusion will commence (91 - 180 min) at 0.35 ng/Kg/min and then increase to 0.70 ng/Kg/min (181- 270 min), a rate which will be maintained till the end of the study (1330).

Study B (0.8mU/Kg/min): Approximately 1-2 weeks after the first study visit, subjects will be asked to return to the CRTU. This study visit will be similar to Study A. However, insulin will be infused at 0.8mU/Kg/min 0 to 270 minutes.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit 15 otherwise healthy subjects using intramural and local extramural advertising after approval from the Mayo Clinic Institutional Review Board. Individuals who express interest in participating will be invited for a screening visit. Individuals with a BMI < 19 or > 28 kg/m2 will be excluded from the study to avoid potential confounding effects that may result from extreme leanness or from obesity. Subjects will have no known systemic illness, taking any medication that could affect glucose metabolism and no history of upper gastrointestinal surgery.

Exclusion Criteria:

* Subjects < 18 years of age or > 40 years of age will not be studied to minimize the potential confounding effects of age on glucagon and insulin action. The subjects will not be taking medications that affect glucose metabolism (to be determined by PI) and have no history of chronic illness or upper gastrointestinal surgery. We are seeking to recruit subjects who do not have diabetes (fasting glucose <100mg/dL).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is a cross-over study - subjects participated in both arms
Groups:
- 0.4 Then 0.8: During the first euglycemic clamp insulin will be infused at 0.4mU/Kg/Min
  Subjects will undergo a 15 day 'withdrawal period'
  During the second euglycemic clamp insulin will be infused at 0.8mU/Kg/Min
- 0.8 Then 0.4: During the euglycemic clamp insulin will be infused at 0.8mU/Kg/Min
  Subjects will undergo a 15 day 'withdrawal period'
  During the second euglycemic clamp insulin will be infused at 0.4mU/Kg/Min
Period: Overall Study
Arm/Group | 0.4 Then 0.8 | 0.8 Then 0.4
Started | 5 | 7
Completed | 5 | 5
Not Completed | 0 | 2
Not completed — IV access lost during the study | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 0.4 Then 0.8: Subjects will undergo the 0.4 clamp first during which insulin is infused at 0.4mU/Kg/Min
  following a suitable washout period,
  Subjects will undergo the 0.8 clamp second during which insulin is infused at 0.8mU/Kg/Min
- 0.8 Then 0.4: Subjects will undergo the 0.8 clamp first during which insulin is infused at 0.8mU/Kg/Min
  following a suitable washout period,
  Subjects will undergo the 0.4 clamp second during which insulin is infused at 0.4mU/Kg/Min
- Total: Total of all reporting groups
Arm/Group | 0.4 Then 0.8 | 0.8 Then 0.4 | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Analysis in people completing both arms
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 5 | 10
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis in people completing both arms
  years
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 34 (13) | 37 (10) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production (EGP)
Description: is calculated by tracer-based measurement and expressed per kg lean body mass
Time Frame: It will be quantified at 90, 180 and 270 minutes for the study with 0.4mU insulin infusion and compared to values obtained for the study with 0.8mU insulin infusion at the same timepoints
Measure: Mean (Standard Error); unit: umol/kg/min
Groups:
- 0.4mU Insulin: During the euglycemic clamp insulin will be infused at 0.4mU/Kg/Min
  0.4mU Insulin: Insulin infused at 0.4 mU/Kg/min
- 0.8mU Insulin: During the euglycemic clamp insulin will be infused at 0.8mU/Kg/Min
  0.8mU Insulin: Insulin infused at 0.8 mU/Kg/min
Arm/Group | 0.4mU Insulin | 0.8mU Insulin
Number analyzed (Participants) | 10 | 10
umol/kg/min
  At 90 minutes | 4.99 (0.53) | 5.02 (0.74)
  At 180 minutes | 6.82 (0.82) | 5.52 (0.96)
  At 270 minutes | 8.48 (1.07) | 5.38 (1.13)

ADVERSE EVENTS:
Time Frame: 3 months
Description: These young healthy participants were in the study for duration of time between screening, and the end of the last experiment. Each of the experiments was 270 minutes long but subjects were admitted the night before and monitored in house till the end of the experiment. After the first experiment there was a 15 day waiting period and then another experiment (with admission the night before).
Groups:
- 0.4 Events: Events occurring during the 0.4 euglycemic clamp when insulin was infused at 0.4mU/Kg/Min
- 0.8 Events: Events occurring during the 0.8 euglycemic clamp when insulin was infused at 0.8mU/Kg/Min
Arm/Group | 0.4 Events | 0.8 Events
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.4 Events (N=12) | 0.8 Events (N=12)
Phlebitis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The main caveat is that during the experiment insulin is kept constant - i.e. not quite like what happens in the postprandial situation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT04461015/Prot_SAP_000.pdf